CLINICAL TRIAL: NCT06140719
Title: A Retrospective and Prospective Observational Sub-Study for Diffuse Midline Glioma and Diffuse Intrinsic Pontine Glioma
Brief Title: xPedite: A Study to Expedite DIPG and DMG Research
Status: Recruiting | Type: Observational
Sponsor: xCures (Industry)
Responsible Party: Sponsor
Other Study IDs: XPED-2023
Record Dates: First submitted 2023-11-07; First posted 2023-11-20 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Oncology; DIPG; DMG
Keywords: DIPG; DMG; Diffuse Midline Glioma; Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Neoplasms; Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will gather data from new and existing patients with patient medical records, and patient/family/caregiver reported information to establish a clear natural history of disease suitable to serve as an external, contemporary or historical control arm for future therapeutic development programs of drugs, devices, or biologic interventions in DMG or DIPG.

DETAILED DESCRIPTION:
xPEDITE is a completely virtual, decentralized, nationwide,real-time, real-world observational study to collect, annotate, standardize, and report the critical data elements of DMG, inclusive of DIPG, in a regulatory-compliant framework. Patients participate by eConsent to the pan-cancer master observational protocol XCELSIOR (NCT03793088). This protocol is a sub-study of XCELSIOR and does not require an additional written consent. Medical records are accessed from institutions directly via eFax or paper fax, online from patient EMR portals, direct from DNA/RNA sequencing and molecular profiling vendors, and via electronic health information exchanges. Medical records are received or converted to electronic/digitized formats (CCDA, FHIR, PDF) and sorted by medical record type (clinic visit, in-patient hospital, out-patient clinic, infusion and out-patient pharmacies, etc.) and made machine-readable to support data annotation, full text searches, and natural language processing (NLP) algorithms to further facilitate feature identification. Data elements are annotated comprehensively and longitudinally from diagnosis to final outcome and include patient level clinical features required to report endpoints in DMG and DIPG clinical trials such as anti-cancer interventions, non-cancer medications, genomics/biomarker results, radiological endpoints, steroid use, vitals, demographics, and locations of care, among others. This study does not require data entry by treating site staff or physicians. Centralized data annotation is completed by xCures remote study staff. Data elements are annotated in a central electronic data capture (EDC) system and coded to Observational Medical Outcomes Partnership (OMOP)-based ontologies (SNOMED, LOINC, ICD-O-3, CTCAE, RxNorm, MedDRA, and others) in one process, permitting standardization of verbatim terms from medical records. Data is collected in a 21 CFR Part 11-compliant EDC system with formal QC/QA process, medical review, and source data verification. Beyond EMR data, raw DICOM images (MRI, CT files) are collected from all sites of care and de-identified. Imaging will be subjected to a blinded central radiological review to assess sizes, and response or progression. For all patients, genomics results (PDFs, variant call files, and raw FASTQ files when available) are collected from commercial and academic sources and centralized. Additionally, patient- and caregiver-reported outcome questionnaires (PROs) are collected to measure the impact of disease and medical care on the patient and family and others living around them to determine the aspects of care that are most important to them. Mobility and neurological assessments will be videoed and submitted at regular intervals to prospectively document changes in clinical status by expert electronic clinician-reported outcomes (ClinROs). Together, these clinical, imaging, biomarker, and assessment data will provide a comprehensive and longitudinal documentation of DMG and DIPG disease course.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of diffuse midline glioma according to the WHO 2021 Classification of Tumors of the Central Nervous System diagnostic criteria including diffuse intrinsic pontine glioma (DIPG). In the absence of a pathologically confirmed diagnosis, a grade IV glioma involving the thalamus, hypothalamus, brainstem, cerebellum, midbrain, or spinal cord, or with a pontine epicenter and diffuse involvement of the pons.
2. Patients with any performance status, comorbidity or disease severity are eligible
3. Patients or their legally-authorized representative must be willing and able to provide electronic, informed consent (and assent, if applicable)
4. Informed consent obtained for the XCELSIOR longitudinal outcomes registry (NCT03793088).
5. Patients must be a resident of or receiving care within the United States or US territories.

Exclusion Criteria:

1. Patient or legally-authorized representative is unable to provide informed consent.
2. Patient or caregiver is unable to complete the PRO and ClinRO by an electronic platform.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 400 patients of any age who have been diagnosed with diffuse midline glioma (DMG) or diffuse intrinsic pontine glioma (DIPG).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 12 months
  OS is defined as time from first dose of treatment to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  ORR is defined as the proportion of patients with a documented complete response (CR) or partial response (PR) as assessed by RANO or RAPNO.
Clinical Benefit Rate (CBR) | 12 months
  CBR defined as the proportion of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) as assessed by RANO or RAPNO

CONTACTS AND LOCATIONS:
Overall Officials: Mark Shapiro, PhD, Principal Investigator — xCures
Locations (1):
- xCures, Inc., Los Altos, California, United States

REFERENCES:
- See also: xCures Website — https://www.xcures.com/patients/